CLINICAL TRIAL: NCT04128449
Title: Modifications in the Anaerob Threshold in Cyclists (DHA)
Brief Title: Modifications in the Anaerob Threshold in Cyclists by Consuming Docosahexaenoic Acid (DHA)
Acronym: MATCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-0004
Record Dates: First submitted 2018-05-15; First posted 2019-10-16 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Performance
Keywords: performance; cyclists; docosahexaenoic acid; anaerobic threshold
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- docosahexaenoic acid (Experimental): 1,66 grams/24 hours (5 dragees)
  Interventions: Dietary Supplement: docosahexaenoic acid
- Placebo (Placebo Comparator): sunflower oil (5 dragees)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: docosahexaenoic acid — 5 dragees every 24 hours
  Arms: docosahexaenoic acid
Dietary Supplement: Placebo — 5 dragees every 24 hours
  Arms: Placebo

SUMMARY:
In a double-blind, parallel randomized clinical trial with 38 cyclists in whom the performance improvement was determined after the consumption of docosahexaenoic acid for one month.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 75 years old.
* Cyclists who train three or four times a week.

Exclusion Criteria:

* Suffering some type of chronic disease.
* Consume habitually pharmacological treatments that could influence the physiological or biochemical responses to be analyzed in the present work.
* Consumption in the month prior to the start of the study, or during the performance of the same, functional food enriched with omega-3 fatty acids.
* To present during the performance of the stress tests, any of the absolute or relative contraindications dictated by the American College of Sports Medicine (ACSM, 1999) 15 would be duly informed and excluded from the present study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
ergospirometry variable: heart rate | The change was evaluated after one month of product consumption.
  It was done with a bicycle with electromagnetic resistance (Spin Trainer ;Technogym). Heart rate was measured in beats per minute.
ergospirometry variable: absolute oxygen consumption | The change was evaluated after one month of consumption of the product
  It was done with a bicycle with electromagnetic resistance (Spin Trainer ;Technogym).It was measured in milliliters per minute

SECONDARY OUTCOMES:
ergospirometry variable:respiratory ratio | The change was evaluated after one month of consumption of the product
  It was done with a bicycle with electromagnetic resistance (Spin Trainer ;Technogym). Through the oxycon pro jaeger gas analyzer.
ergospirometry variable: oxygen equivalent | The change was evaluated after one month of consumption of the product
  It was done with a bicycle with electromagnetic resistance (Spin Trainer ;Technogym). Through the oxycon pro jaeger gas analyzer.
blood variables: Natremia, potassium, chloremia, calcemia, , bicarbononatemia, ph, lactacidemia. | The change was evaluated after one month of product consumption.
  The following variables were analyzed: The variables are analyzed using the ABL 77 radiometer. The unit of measurement is mmol / L.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain